CLINICAL TRIAL: NCT05115968
Title: Single Cell Sequencing to Examine the Pathogenesis of Adenotonsillar Hypertrophy in Children With Obstructive Sleep Apnoea
Brief Title: Single Cell Sequencing of Tonsillar Tissue in Children With OSA
Status: Recruiting | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Kate Ching Ching Chan, Clinical Professional Consultant, Chinese University of Hong Kong
Other Study IDs: SCSAT_protocol_version 1.0
Record Dates: First submitted 2021-09-22; First posted 2021-11-10 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Obstructive Sleep Apnea of Child
MeSH Terms: interventions — Tonsillectomy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Tonsillar tissue
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- OSA case: Chinese children aged 6-11 years old with habitual snoring (≥3 nights per week) and polysomnography (PSG) confirmed OSA (obstructive apnoea hypopnoea index (OAHI) of ≥1/hour), with adenotonsillar hypertrophy and clinical indications for adenotonsillectomy will be recruited as cases.
  Interventions: Procedure: Tonsillectomy
- Control: Non-OSA subjects (with PSG OAHI <1/hour) who undergo adenotonsillectomy for other reasons such as recurrent tonsillitis.
  Interventions: Procedure: Tonsillectomy

INTERVENTIONS:
Procedure: Tonsillectomy — Subjects who are diagnosed to have OSA with adeontonsillar enlargement will undergo adenotonsillectomy if it is clinically indicated. Adenotonsillar tissue will be obtained for single cell sequencing. Controls will be non-OSA subjects (with PSG OAHI <1/hour) who undergo adenotonsillectomy for other reasons such as recurrent tonsillitis.

SUMMARY:
Obstructive sleep apnoea (OSA) in children is a prevalent sleep disorder, and is characterised by repetitive complete or partial upper airway obstruction during sleep. It is an important disease as it is associated with a large spectrum of end-organ morbidities.

Adenotonsillar hypertrophy is the commonest cause of OSA in children, however, the cause of the lymphoid tissue hypertrophy in some individuals but not the others remains unknown. To address the cellular heterogeneity and immune cell involvement in adenotonsillar hypertrophy, here, we propose to employ single-cell sequencing analysis to identify the cell-specific expression patterns associated with the disease, which will enhance our understanding of the pathogenesis of tonsillar hypertrophy in children with OSA and may provide directions for development of novel therapy.

ELIGIBILITY:
Inclusion Criteria:

Case: Chinese children aged 6-11 years old with habitual snoring (≥3 nights per week) and polysomnography (PSG) confirmed OSA (obstructive apnoea hypopnoea index (OAHI) of ≥1/hour), with adenotonsillar hypertrophy and clinical indications for adenotonsillectomy will be recruited as cases.

Control: Non-OSA subjects (with PSG OAHI <1/hour) who undergo adenotonsillectomy for other reasons such as recurrent tonsillitis.

Exclusion Criteria:

Previous upper airway surgery, genetic or syndromal disease, congenital or acquired neuromuscular disease, congenital or acquired immunodeficiency, known metabolic syndrome, craniofacial abnormalities.

Ages: 6 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Case: Chinese children aged 6-11 years old with habitual snoring (≥3 nights per week) and polysomnography (PSG) confirmed OSA (obstructive apnoea hypopnoea index (OAHI) of ≥1/hour), with adenotonsillar hypertrophy and clinical indications for adenotonsillectomy will be recruited as cases.
  Control: Non-OSA subjects (with PSG OAHI <1/hour) who undergo adenotonsillectomy for other reasons such as recurrent tonsillitis.
Sampling Method: Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Tonsil cell characteristics | Through study completion, an average of 2 years
  Cells characteristics by single-cell sequencing of the adenotonsillar tissue in children with OSA.

CONTACTS AND LOCATIONS:
Overall Officials: Kate C Chan, MBChB, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Prince of Wales Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No